CLINICAL TRIAL: NCT01652053
Title: A Pilot Clinical Study to Assess the Safety and Effectiveness of the InterCushion Disc Nucleus Prosthesis in Patients Receiving Discectomy
Brief Title: A Pilot Study of the InterCushion Disc Nucleus Prosthesis (DNP) in Patients Receiving Discectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vertebral Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP 2010-001
Record Dates: First submitted 2012-07-24; First posted 2012-07-27 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Disk, Herniated
Keywords: InterCushion
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Disc Nucleus Replacement: Disc Nucleus Replacement (InterCushion DNP)
  Interventions: Device: Disc Nucleus Replacement (InterCushion DNP)

INTERVENTIONS:
Device: Disc Nucleus Replacement (InterCushion DNP) — The device is intended for spinal arthroplasty in skeletally mature patients with leg pain due to a herniated disc with or without back pain, who are having a discectomy at one level from L2 -S1. These patients should have no spondylolisthesis at the involved level.
  Other Names: InterCushion Disc Nucleus Prosthesis (DNP)

SUMMARY:
The primary endpoints of the investigation will include assessment of the maintenance of disc height demonstrated by radiographic evidence based on plain radiographs and MRI and relief of pain as measured by Visual Analog Scale (VAS) at six months post-surgery. It is anticipated that outcomes with the InterCushion Disc Nucleus Prosthesis (DNP) will be comparable to or better than the historical published results for discectomy alone.

DETAILED DESCRIPTION:
All patients will be followed for at least 24 months once enrolled in the study. Clinical evaluations will be conducted before surgery (baseline), intraoperative, 2 week (± 1 week), 6 week (± 1 week), 3 months (± 2 weeks), 6 months (± 1 month), 12 months (± 2 months) and 24 months (± 2 months).

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed and dated a study specific informed consent form approved by the reviewing Institutional Review Board or Ethics Committee.
* Patient is 21 to 60 years of age.
* Patient is skeletally mature
* Patient requires a discectomy of one level from L2-S1.
* Patient has less than 50% loss of disc height at the affected level.
* Patient has persistent pain (predominantly leg pain, although some back pain that occurred at the same time as the leg pain and is believed to be associated with the disc herniation will not disqualify the patient from participating in this study) and symptoms despite a minimum of six weeks of non-operative treatment.
* Patient X-ray, CT or MR evidence of a herniated disc at the affected level.
* Patient has a minimum leg pain score of 6 cm on a 10 cm (i.e. 60 mm on a 100 mm) point visual analog scale (VAS).
* Patient has a minimum Oswestry Disability Index score of 40% (based upon a 100% scale).
* Patient is physically and mentally willing and able to comply with the postoperative scheduled clinical and radiographic evaluations and rehabilitation.

Exclusion Criteria:

* Patient has had any previous surgery at the affected levels.
* Patient has had any attempt at spinal fusion, at any lumbar levels.
* Patient has motion of < 3 degrees on pre-operative lateral flexion/extension radiographs
* Patient has a BMI
* Patient has severe osteoporosis of the spine.
* Patient has previously undergone chemotherapy, immunosuppressive therapy or radiation to the local area.
* Patient has active local or systemic infection.
* Patient has any known active malignancy.
* Patient has rheumatoid arthritis or systemic lupus erythematosus, or other chronic, inflammatory autoimmune disorder.
* Patient has ankylosing spondylitis or other spondyloarthropathy.
* Patient has spondylolisthesis.
* Patient is pregnant or plans to become pregnant during the course of the study.
* Patient has other concurrent physical or mental conditions that are likely to affect their outcome.
* Patient has congenital stenosis
* Patient is diabetic.
* The patient has osteoporosis or severe osteopenia as determined by the Investigator. Females over 40 with bone density score less than -1. A clinical SCORE calculator may also be utilized for females over 40 years of age.
* Patient has significant facet disease.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The protocol includes skeletally mature patients, both male and female, 18 to 60 years old suffering from a herniated disc (confirmed by X-ray, CT or MRI) with persistent leg pain.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Decrease in ODI | 6 months
  Improvement in the Oswestry Disability Index (ODI) score i.e. decrease of 15% or better ODI.
Decrease in VAS | 6 months
  Improvement in leg pain evidenced by decrease in pain score of at least 2 cm (i.e. 20 mm) on the visual analog scale (VAS)
Maintenance of post-operative disc height | 6 months
  Disc at the treated level is collapsed by ≤ 15% when compared to an adjacent health level.
Mobility of treated segment | 6 months
  Motion of ≥ 3 degrees on lateral flexion/extension radiographs
Neurologic deficits | 6 months
  No new permanent neurological deficit or worsening of an existing permanent neurological deficit

SECONDARY OUTCOMES:
Maintenance or decrease in ODI | 12 and 24 months
  Maintenance of improvement or further improvement in the Oswestry Disability Index (ODI) score measured at six months i.e. decrease of 15% or better ODI.
Maintenance or decrease in VAS | 12 and 24 months
  Maintenance of improvement or further improvement in leg pain evidenced by decrease in pain score on the visual analog scale (VAS)
Maintenance of post-operative disc height. | 12 and 24 months
  Disc at the treated level is collapsed by ≤ 15% when compared to an adjacent health level.
Mobility of treated segment | 12 and 24 months
  Motion of ≥ 3 degrees on lateral flexion/extension radiographs
Neurological deficits | 12 and 24 months
  No new permanent neurological deficit or worsening of an existing permanent neurological deficit

OTHER OUTCOMES:
Failures | 6, 12 and 24 months
  Revision: is a procedure that adjusts or in any way modifies or removes part of the original implant configuration, with or without replacement of a component.
  Removal: is a procedure where the entire original system configuration is removed with or without replacement.
  Supplemental fixation: a procedure in which additional instrumentation not under study is implanted.

CONTACTS AND LOCATIONS:
Overall Officials: Phillip F de Muelanaere, MD, Principal Investigator — Brandon General Hospital
Locations (1):
- Brandon Regional Health Center, Brandon, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No